CLINICAL TRIAL: NCT01644487
Title: Efficacy of Self-Expanding Nitinol Stent Versus Balloon Angioplasty Alone for the Below The Knee Arteries Following Successful Balloon Angioplasty Trial (Korean Vascular Intervention Multicenter Study)
Brief Title: Self-Expanding Nitinol Stent Versus Balloon Angioplasty Alone for the Below The Knee Arteries(SENS-BTK)
Acronym: SENS-BTK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Korea University Guro Hospital (Other)
Responsible Party: Principal Investigator, Seung Woon Rha, Professor, Korea University Guro Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EV-10302
Record Dates: First submitted 2012-07-17; First posted 2012-07-19 (Estimated); Last update posted 2019-08-14 (Actual); Status verified 2017-08

CONDITIONS: Critical Limb Ischemia; Infrapopliteal Arterial Occlusive Disease
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia | interventions — Angioplasty, Balloon

STUDY DESIGN:
Intervention Model Description: Provisional stenting with SMART(n=173), Provisional stenting with Complete SE(n=173)

ARMS (2):
- Primary stenting (Experimental): A group of patients who will undergo subsequent primary stenting following successful conventional balloon angioplasty
  Interventions: Device: self-expanding nitinol stent
- Balloon only (Active Comparator): A group of patients who will undergo routine conventional balloon angioplasty alone without stenting
  Interventions: Device: balloon angioplasty

INTERVENTIONS:
Device: self-expanding nitinol stent — A group of patients who will undergo subsequent primary stenting following successful conventional balloon angioplasty
  Other Names: Xpert stent
  Arms: Primary stenting
Device: balloon angioplasty — A group of patients who will undergo routine conventional balloon angioplasty alone without stenting
  Arms: Balloon only

SUMMARY:
The objectives of this study are to compare directly conventional balloon angioplasty alone versus. balloon angioplasty with routine stenting - that is, to determine whether angioplasty with self-expanding stent is superior to conventional balloon angioplasty - in the infrapopliteal arterial occlusive lesions of critical limb ischemia patients by collecting and analyzing the cases of each patient group in a prospective multicenter randomized clinical trial, and to clarify main factors affecting mid- and long-term clinical effects of angioplasty with self-expanding stent in the infrapopliteal arteries.

Hypothesis: Balloon PTA followed by routine stenting with self-expanding nitinol stent in critical limb ischemia patients with infrapopliteal arterial occlusive lesions is superior to conventional PTA in the aspect of vascular restenosis rate.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic critical limb ischemia (Rutherford 4 - 6)
* Patients with signed informed consent
* Target lesion length < 8 cm by angiographic estimation
* Stenosis of >50% or occlusive atherosclerotic lesion of the ipsilateral infrapopliteal artery
* Reference vessel diameter should be 2.0-4.5 mm

Exclusion Criteria:

* Patient has a known allergy to heparin, aspirin, or other anticoagulant/antiplatelet therapies or a bleeding diatheses or is unable, or unwilling, to tolerate such therapies
* Patient takes warfarin
* Patient has a history of previous life-threatening contrast media reaction
* Patient is currently enrolled in another investigational device or drug trial
* Patient is currently breast-feeding, is pregnant, or intends to become pregnant
* Patient is mentally ill or retarded
* Acute critical limb ischemia
* Major bleeding history within prior 2 months
* Severe hepatic dysfunction (> 3 times normal reference values)
* Significant leucopenia, neutropenia, thrombocytopenia, anemia, or known bleeding diathesis
* Life expectancy <1 year due to comorbidity
* Reference segment diameter is not suitable for available stent design
* Previously implanted stent(s) or PTA at the same lesion site
* Inflow-limiting arterial lesions left untreated

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2012-07; Primary Completion 2016-09-06 (Actual); Study Completion 2018-10-10 (Actual)

PRIMARY OUTCOMES:
Angiographic binary restenosis rate | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Guro Hospital, Seoul, South Korea